CLINICAL TRIAL: NCT05627856
Title: An Open, Multicenter, Phase Ib/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics/Pharmacokinetics, and Antitumor Activity of GNC-038 Injection in Relapsed or Refractory NK/ T-cell Lymphoma, AITL, and Other NHL
Brief Title: A Study of GNC-038 Injection in Patients With Relapsed or Refractory NK/ T-cell Lymphoma, AITL, and Other NHL
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: SystImmune Inc. (Industry); Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GNC-038-105
Record Dates: First submitted 2022-11-08; First posted 2022-11-28 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: NK/T Cell Lymphoma; Vascular Immunomother T Cell Lymphoma; Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study treatment (Experimental): Participants receive GNC-038 as intravenous infusion for the first cycle (2 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: GNC-038

INTERVENTIONS:
Drug: GNC-038 — Administration by intravenous infusion

SUMMARY:
To explore the safety and efficacy of GNC-038 in relapsed or refractory NK/T cell lymphoma, vascular immunomother T cell lymphoma, and other relapsed or refractory NHL, and to determine MTD, MAD, DLT, and RP2D of GNC-038, as well as its pharmacokinetic characteristics and immunogenicity.

DETAILED DESCRIPTION:
Phase Ib: To explore the safety and preliminary effectiveness of GNC-038 under the administration mode of "intravenous infusion for 2h to 4h, once a week (IV, QW), 2 weeks as one cycle", and to determine MTD, MAD, DLT and RP2D of GNC-038. The pharmacokinetic characteristics and immunogenicity of GNC-038 will be evaluated. Phase II: To explore the efficacy, safety and tolerability, pharmacokinetic characteristics and immunogenicity of GNC-038.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects can understand the informed consent, voluntarily participate in and sign the informed consent.
2. No gender restriction.
3. Age: ≥18 and ≤75 years old.
4. Expected survival time ≥3 months.
5. Patients with histologically confirmed NK/T cell lymphoma or vascular immunomother T cell lymphoma.
6. Patients with relapsed/refractory NK/T cell lymphoma (R/R NKTCL) or relapsed/refractory vascular immunomother T cell lymphoma (AITL):

1) Patients with recurrent or refractory vascular immunomother T cell lymphoma after initial treatment.

2) Patients with NK/T cell lymphoma need to have received systematic therapy with asparaginase regimen in the past, and have received radiotherapy for single lesion recurrence or refractory treatment.

Difficult-to-treat definition: i) the curative effect of end-line treatment did not reach PR; Or ii) disease progression within 6 months after terminal line treatment.

7. In the screening period, there were measurable lesions (lymph node lesions with any length ≥1.5cm or exodal lesions with any length > 1.0cm, all of which had metabolic activity).

8. Physical status score ECOG ≤2 points. 9. The adverse reactions of previous antitumor therapy were restored to CTCAE level 5.0 evaluation ≤ level 1 (except for indicators that the researchers considered might be related to the disease, such as anemia, and toxicities that the researchers judged to have no safety risk, such as hair loss, grade 2 peripheral neurotoxicity, stable hypothyroidism after hormone replacement therapy, etc.).

10. Organ function level before initial administration meets the following requirements: Bone marrow function: without blood transfusion within 7 days prior to screening, without G-CSF (without long-acting rising white needle within 2 weeks) and drug correction: Absolute neutrophil count (ANC) ≥1.0×109/L (≥0.5×109/L for subjects with bone marrow infiltration); Hemoglobin ≥80 g/L (≥70g/L for subjects with bone marrow infiltration); Platelet count ≥75×109/L; Liver function: total bilirubin ≤1.5 ULN (Gilbert's syndrome ≤3 ULN), transaminase (AST/ALT) ≤2.5 ULN (subjects with liver tumor invasive changes ≤5.0 ULN) within 7 days before screening without liver protection drugs; Renal function: creatinine (Cr) ≤1.5 ULN and creatinine clearance (Ccr) ≥50 ml/min (according to Cockcroft and Gault formula); Urine routine /24 hours urine protein quantification: qualitative urine protein ≤1+ (if qualitative urine protein ≥2+, 24 hours urine protein < 1g can be included in the group); Cardiac function: left ventricular ejection fraction ≥50%; Coagulation function: fibrinogen ≥1.5g/L; Activated partial thrombin time (APTT) ≤1.5 ULN; Prothrombin time (PT) ≤1.5 ULN.

11. Fertile female subjects or fertile male subjects with partners must use highly effective contraception from 7 days prior to the first dose until 12 weeks after termination of treatment. A fertile female subject must have a negative serum/urine pregnancy test within 7 days prior to initial dosing.

12. Subject is able and willing to comply with visits, treatment plans, laboratory tests, and other study-related procedures as specified in the study protocol.

Exclusion Criteria:

1. According to NCI-CTCAE v5.0, it was defined as ≥ grade 3 pulmonary disease; Patients who currently have interstitial lung disease (ILD) (except those who previously had interstitial pneumonia and have recovered).
2. Active infections requiring systemic treatment, such as severe pneumonia, bacteremia, sepsis, etc.
3. Active tuberculosis.
4. Patients with hemophagocytic syndrome.
5. Patients with lesions invading pulmonary great vessels.
6. Active patients with autoimmune diseases, such as: systemic lupus erythematosus, systemic treatment of psoriasis, rheumatoid arthritis, inflammatory bowel disease, and hashimoto's thyroiditis, etc., with the exception of type I diabetes, only replacement therapy can control the hypothyroidism, no systemic treatment of skin disease (e.g., vitiligo, psoriasis), B cells caused by autoimmune disease.
7. Non-melanoma skin cancer in situ, superficial bladder cancer in situ, cervical cancer in situ, gastrointestinal intramucosal cancer, breast cancer, localized prostate cancer and other malignant tumors that were combined with other malignant tumors within 5 years prior to the first administration of the drug, except those that the researchers thought could be included.
8. HBsAg positive or HBcAb positive, and HBV-DNA detection ≥ detection value lower limit (HBV-DNA detection in the normal range and regular use of anti-HBV drugs except patients); HCV antibody was positive and HCV-RNA≥ lower limit of detection value.
9. Poorly controlled hypertension (systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg).
10. A history of severe cardiovascular and cerebrovascular diseases, including but not limited to:

    Severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias and degree III atrioventricular block that require clinical intervention; Prolonged QT interval at rest (QTc > 450 msec in men or 470 msec in women); Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other grade 3 or higher cardiovascular and cerebrovascular events occurring within 6 months prior to initial administration; Present with heart failure ≥II on the New York Heart Association (NYHA) cardiac function scale.
11. Patients with a history of allergy to recombinant humanized antibodies or to any excipient component of GNC-038.
12. Pregnant or breastfeeding women.
13. Patients with central nervous system invasion.
14. Patients who received major surgery within 28 days prior to drug administration in this study, or planned to undergo major surgery during the study period (except for procedures such as puncture or lymph node biopsy).
15. Previous recipients of organ transplantation or allogeneic hematopoietic stem cell transplantation (Allo-HSCT).
16. Autologous hematopoietic stem cell transplantation (Auto-HSCT) within 24 weeks before starting GNC-038 therapy.
17. Immunosuppressants are being used, including, but not limited to, cyclosporine, tacrolimus, etc. within 2 weeks prior to treatment with GNC-038.
18. Radiotherapy was received within 4 weeks prior to the initiation of GNC-038 therapy.
19. Received chemotherapy and small molecule targeted therapy within 2 weeks prior to treatment.
20. Received CAR-T therapy within 12 weeks prior to initiation of GNC-038 therapy.
21. Participants in any other clinical trial within 4 weeks prior to administration of this trial.
22. A history of immunodeficiency, including HIV positive testing, or other acquired, congenital immunodeficiency diseases.
23. Other conditions deemed unsuitable for participation in this clinical trial by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Phase Ib: Dose Limited Toxicity (DLT) | Up to 16 days after the first dose
  The incidence and severity of adverse events (TEAE) during treatment were graded according to the National Cancer Institute Standard for Common Terminology for Adverse Events (NCI-CTCAE, v5.0).
Phase Ib: Maximum Tolerated dose (MTD) or maximum administered dose (MAD) | Up to 16 days after the first dose
  In the dose increment stage, the highest dose whose estimated DLT rate is closest to the target DLT rate but does not exceed the upper bound of the equivalent interval of DLT rate is selected as MTD.
Phase Ib: Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of GNC-038. The type, frequency and severity of TEAE will be evaluated during the treatment of GNC-038.
Phase Ib: Recommended Phase II Dose (RP2D) | Up to 16 days after the first dose
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of GNC-038.
Phase II: Objective response rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.

SECONDARY OUTCOMES:
Phase Ib: Objective response rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
Phase Ib: Progression-free survival (PFS) | Up to approximately 24 months
  The PFS is defined as the time from the participant's first dose of GNC-038 to the first date of either disease progression or death, whichever occurs first.
Phase Ib: Disease control rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Phase Ib:Duration of response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Phase Ib: Complete Response (CR) | Up to approximately 24 months
  Disappearance of all target lesions.
Phase Ib: Adverse Events of Special Interest (AESI) | Up to approximately 24 months
  AESI is an event of scientific and medical interest specific to the sponsor's product or research project.
Phase Ib: Cmax | Up to 16 days after the first dose
  Maximum serum concentration (Cmax) of GNC-038 will be investigated.
Phase Ib:Tmax | Up to 16 days after the first dose
  Time to maximum serum concentration (Tmax) of GNC-038 will be investigated.
Phase Ib:AUC0-inf | Up to 16 days after the first dose
  Blood concentration - Area under time line.
Phase Ib: AUC0-T | Up to 16 days after the first dose
  Blood concentration - Area under time line.
Phase Ib: CL(Clearance) | Up to 16 days after the first dose
  To study the serum clearance rate of GNC-038 per unit time.
Phase Ib: T1/2 | Up to 16 days after the first dose
  Half-life (T1/2) of GNC-038 will be investigated.
Phase Ib: Anti-drug antibody (ADA) | Up to approximately 24 months
  Frequency and titer of anti-GNC-038 antibody (ADA) will be evaluated.
Phase II: Progression-free survival (PFS) | Up to approximately 24 months
  The PFS is defined as the time from the participant's first dose of GNC-038 to the first date of either disease progression or death, whichever occurs first.
Phase II: Disease control rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Phase II:Duration of response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Phase II: Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of GNC-038. The type, frequency and severity of TEAE will be evaluated during the treatment of GNC-038.

CONTACTS AND LOCATIONS:
Overall Officials: Wenyu Li, PHD, Principal Investigator — Guangdong Provincial People's Hospital; Huiqiang Huang, PHD, Principal Investigator — Sun Yat-sen University
Locations (2):
- China (2):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong